CLINICAL TRIAL: NCT04108923
Title: Comparative Study Between Ligasure Versus Conventional Vessel Ligation in Thyroidectomy " Randomised Controlled Study"
Brief Title: Comparative Study Between Ligasure Versus Conventional Vessel Ligation in Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abadeer Raafat Marsis Rizallah, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemostasis in thyroidectomy
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Thyroid Diseases
Keywords: Thyroidectomy; Ligasure; Vessel ligation
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligasure ( group A) (Active Comparator)
  Interventions: Device: Ligasure
- Conventional vessel ligation (group B) (Active Comparator)
  Interventions: Procedure: Conventional vessel ligation

INTERVENTIONS:
Device: Ligasure — the vessel sealing device ( ligasure covidien ) which seals vessels by fusing the inner layers of the vessel wall
  Arms: Ligasure ( group A)
Procedure: Conventional vessel ligation — Conventional vessel ligation either tying and /or clipping of blood vessels
  Arms: Conventional vessel ligation (group B)

SUMMARY:
To compare between ligasure versus conventional vessel ligation in thyroidectomy as regards intraoperative and post operative complications rate

DETAILED DESCRIPTION:
The significant vascularity of the thyroid gland and the relatively small operative field makes meticulous hemostasis an important prerequisite in thyroid surgery for successful outcome. The mainstay for achieving hemostasis in thyroidectomy is tying and / or clipping of blood vessels. New technologies have been introduced , among them the vessel sealing device ( ligasure ) which seals vessels by fusing the inner layers of the vessel wall with minimal levels of thermal dispersion burning and tissue friction thereby reducing incidence of accidental burns . This study is designed to evaluate the safety and efficacy of using ligasure compared with conventional vessel ligation in open thyroid surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient who will undergo lobectomy , subtotal thyroidectomy , total thyroidectomy at time of study
* Any age

Exclusion Criteria:

* patient undergoing re-do surgery " completion thyroidectomy "
* patient undergoing concomitant procedures as cervical lymphadenectomy or parathyroidectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Baseline
  Measuring intraoperative blood loss using surgical towels and contents of suction.
  Intraoperatively from skin incision " start of operation " to skin closure "complete the operation "
Post-operative blood loss | From skin closure until one week post operatively
  Measuring postoperative blood loss by measuring contents of drains
Post-operative complications | Postoperatively from day of surgery until one week post operatively
  Including RLN palsy , hypocalcemia , hemorrhage wound infection
Operation time | Baseline
  From skin incision to skin closure

SECONDARY OUTCOMES:
Length of hospital stay | Baseline up to two weeks
  Measuring number of days of patient stay in hospital to be pain- free return to activity and work.
  From day of surgery until discharge

REFERENCES:
- [Background] Youssef T, Mahdy T, Farid M, Latif AA. Thyroid surgery: use of the LigaSure Vessel Sealing System versus conventional knot tying. Int J Surg. 2008 Aug;6(4):323-7. doi: 10.1016/j.ijsu.2008.05.005. Epub 2008 May 23. PMID 18585113
- [Background] Vidal O, Saavedra-Perez D, Valentini M, Astudillo E, Fernandez-Cruz L, Garcia-Valdecasas JC. Surgical outcomes of total thyroidectomy using the LigaSure Small Jaw versus LigaSure Precise: A retrospective study of 2000 consecutive patients. Int J Surg. 2017 Jan;37:8-12. doi: 10.1016/j.ijsu.2016.08.241. Epub 2016 Aug 23. PMID 27565244
- [Background] Luo Y, Li X, Dong J, Sun W. A comparison of surgical outcomes and complications between hemostatic devices for thyroid surgery: a network meta-analysis. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1269-1278. doi: 10.1007/s00405-016-4190-3. Epub 2016 Aug 1. PMID 27481528
- [Background] Peker K, Dumanli Ozcan AT, Sahin M, Inal A, Kilic K, Ozcicek F. A comparison of total thyroidectomies carried out through LigaSure and Harmonic Scalpel: a retrospective study. Turk J Med Sci. 2014;44(2):255-60. doi: 10.3906/sag-1210-94. PMID 25536733